CLINICAL TRIAL: NCT01883297
Title: Phase I Study Evaluating the Feasibility and Safety of Infusion of "Re-Stimulated" Autologous TILs Followed by Low-Dose IL-2 Therapy in Patients with Platinum Resistant High Grade Serous Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: "Re-Stimulated" TILs and IL-2 Therapy for Platinum Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILs-001-DC
Record Dates: First submitted 2013-06-11; First posted 2013-06-21 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Recurrent; Platinum-resistant; High Grade Serous Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Measurable; Recurrent; Platinum resistant; Tumor-Infiltrating Lymphocytes; Low-Dose Interleukin-2; Autologous dendritic cells; Anti-CD3 monoclonal antibody; High grade serous ovarian cancer; Fallopian tube cancer; Primary peritoneal cancer; Cyclophosphamide
MeSH Terms: conditions — Recurrence; Fallopian Tube Neoplasms | interventions — Interleukin-2; aldesleukin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Re-Stimulated Tumor-Infiltrating Lymphocytes and interleukin-2 (Experimental): Cyclophosphamide will be given prior to Re-Stimulated Tumor-Infiltrating Lymphocytes, and interleukin-2.
  Interventions: Biological: Re-stimulated tumor-infiltrating lymphocytes (TILs); Biological: Interleukin-2; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Re-stimulated tumor-infiltrating lymphocytes (TILs) — Intravenous infusions: Dose level 1 (3 patients): 3x10^7 TILs (with maximum 3x10^6 autologous dendritic cells); Dose level 2 (3 patients): 1x10^8 TILs (with maximum 1x10^7 autologous dendritic cells); Dose level 3 (3 patients): 3x10^8 TILs (with maximum 3x10^8 autologous dendritic cells)
Biological: Interleukin-2 — Subcutaneous injections of IL-2 x 4 days during the first week and x 5 days the second week with 2 days of rest in between each week of dosing
  Other Names: Aldesleukin, Proleukin, Recombinant Human Interleukin 2
Drug: Cyclophosphamide — Intravenous infusion: 30 mg/kg/day for 2 days (Day -3 and -2 prior to infusion of TILs)
  Other Names: Procytox

SUMMARY:
This is a phase I clinical study for patients with platinum-resistant high grade serous ovarian, fallopian tube, or primary peritoneal cancer, and the response to a combination of cyclophosphamide, autologous tumor-infiltrating lymphocytes (TILs), autologous dendritic cells (DCs), and OKT3 (anti-CD3 antibody), along with low-dose interleukin-2 (IL-2) therapy.

DETAILED DESCRIPTION:
This is a phase I clinical study for patients with platinum-resistant (does not respond to platinum-based chemotherapy) high grade serous ovarian, fallopian tube, or primary peritoneal cancer. Prior to the main treatment, patients will receive cyclophosphamide by vein. Patients will then receive an infusion (given by vein) of autologous tumor-infiltrating lymphocytes (TILs) which will first be taken from the patient, then be stimulated with certain substances called autologous dendritic cells (DCs) and OKT3 (anti-CD3 antibody), and then given back to the patient as an infusion. This is believed to make the TILs work better. TILs are a type of white blood cells that recognizes tumor cells and enter them which causes the tumor cells to break down. After infusion of TILs, low-dose interleukin-2 (IL-2) therapy will be given.

ELIGIBILITY:
Inclusion Criteria (Eligibility for TIL Evaluation):

1. Platinum resistant high grade serous ovarian, fallopian tube, or primary peritoneal cancer.
2. Tumor is suitable for harvest (i.e., lesion to be harvested for TIL evaluation has a total volume of ≥1cm3) or patient has previously undergone tumor harvest under other REB approved studies involving clinical evaluation of TILs.
3. If tumor harvest is required, subject must be a suitable surgical candidate in the opinion of the operating surgeon.
4. Patient age: ≥ 18 years.
5. Clinical performance status of ECOG 0 or 1.
6. Life expectancy > 5 months from the date of consent for TIL evaluation.
7. Ability to understand and has signed the Pre-Screening Consent Form.
8. Patients are willing to be tested for transmissible diseases (active Hepatitis B (HBV) or Hepatitis C (HCV), human immunodeficiency virus (HIV), Human T-Cell Lymphotropic Virus (HTLV), Herpes Simplex Virus (HSV), Cytomegalovirus (CMV), Syphilis (with West Nile Virus only tested between May 1st and November 30th)
9. Confirmation that the Translational Immunotherapy Lab is able to process the specimen
10. If there is a history of allergy to penicillin, gentamycin, streptomycin, or anti-fungals, the ability to generate TILs should first be confirmed with the cell manufacturing lab (i.e., Translational Immunotherapy Laboratory).

Inclusion Criteria (Eligibility for Treatment):

1. Prior to the performance of any study-specific procedure, the subject has signed and dated the informed consent form, approved by a Research Ethics Board (REB), after the nature of the study has been explained and the subject has had the opportunity to ask questions.
2. Recurrent platinum resistant high grade serous ovarian, fallopian tube, or primary peritoneal cancer, with evidence of disease progression from previous line of treatment.
3. Measurable disease by RECIST 1.1.
4. Subjects should have no brain metastases. Note if brain metastases are present, these lesions must undergo definitive treatment with surgery and/or radiation at least 30 days prior to the first dose of lymphodepleting chemotherapy. If in the opinion of the PI or his designee the lesion(s) no longer represents active disease, the subject will be considered eligible.
5. Clinical performance status of ECOG 0 or 1.
6. Life expectancy > 3 months from the date of consent for TIL treatment.
7. Laboratory analyses of tumor-infiltrating lymphocytes (TILs) from the subject must demonstrate that the TILs are suitable for use in protocol treatment (performed by the Translational Immunotherapy Laboratory, Princess Margaret Cancer Centre)
8. More than 30 days has elapsed since any prior systemic therapy at the time of the cell infusion. All subjects' toxicities must have recovered to a CTCAE grade 1 or less; however, patients with residual CTCAE grade 2 neuropathy from previous carboplatin/taxol treatment will not be excluded. Subjects may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to CTCAE grade 1 or less or as specified in the inclusion criteria listed above.
9. Adequate organ function as defined by the following criteria:

   1. Serum ALT ≤ 2.5 x upper limit of normal (ULN) (for patients with liver metastases, serum ALT ≤ 3 x ULN;
   2. Serum AST ≤ 2.5 x upper limit of normal (ULN) (for patients with liver metastases, serum AST ≤ 3 x ULN;
   3. Total serum bilirubin ≤ 2xULN (patients with Gilbert's Syndrome - direct serum bilirubin ≤ 2 x ULN);
   4. Absolute neutrophil count (ANC) ≥ 1.5x109/L;
   5. Platelets ≥100x109/L;
   6. Hemoglobin ≥ 90 g/L for female;
   7. Alkaline phosphatase ≤ 2 x ULN;
   8. Serum creatinine within normal institutional limits OR serum creatinine clearance ≥ 60 mL/min/1.73m2 for patients with creatinine levels above institutional normal;
   9. Serum lipase≤ 1.5 x ULN;
   10. Serum amylase ≤ 1.5 x ULN
10. Women of child-bearing potential must have a negative pregnancy test. Acceptable birth control failure rate of less than or equal to 1% when used consistently and correctly such as implants, injectables, combined oral contraceptives, double barrier, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner. Subjects are considered to be not of child bearing potential if they are considered to be post-menopausal or surgically sterilized (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy. Women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, ovarian suppression or any other reversible reason.

Exclusion Criteria:

1. Subjects with ongoing or prior use systemic steroid therapy within 4 weeks before the TILs infusion will be excluded. Use of topical, intranasal and inhaled corticosteroids, or systemic corticosteroids at physiologic doses are allowed. Oral steroid use as premedication to prevent allergic reactions to radiologic contrast is allowed.
2. Subjects cannot be HIV positive.
3. Subjects cannot have active hepatitis B or hepatitis C, syphilis, or Human T-Cell Lymphotropic Virus (HTLV).
4. The number of prior lines of chemotherapy is not limited. However, if the subject has had ≥3 lines of prior chemotherapy for platinum refractory or platinum resistant disease, documentation of a response to one of these lines is required. Response can be defined by RECIST 1.1 or CA125 as defined by the modified GCIG criteria (See Section 11).
5. The subject cannot have any active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, uncontrolled psychiatric disorders, or other conditions that may affect compliance with the trial.
6. The subject must have no active underlying cardiac illnesses defined by positive stress test, LVEF<40% or ongoing life-threatening arrhythmias (i.e., for patients older than 60 years of age or otherwise clinically indicated).
7. Subjects who have a prolonged history of cigarette smoking or symptoms of respiratory dysfunction will be excluded if they have an abnormal pulmonary function test as evidenced by a FEV1 < 60% predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-01; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of occurrences and severity of side effects | Starting at first dose of study treatment up to 10 years
  Toxicities will be monitored on an ongoing basis by the investigators. Toxic effects will be categorized using the CTCAE v4.0 and will be reported using summary statistics. The highest toxicity for each patient in each category or subcategory will be described. Both events related and unrelated to treatment will be captured. The total number of episodes for each event reported, the severity and attribution to study therapy of each episode reported will also be displayed.

SECONDARY OUTCOMES:
Clinical response to treatment | 6 weeks after treatment
  Evaluation of the clinical response (clinical tumor regression), which will be monitored and reported according to RECIST v1.1 criteria and Immune-Related Response Criteria.
Number of patients with an immunity and no immunity to the study treatment | From start of the study up to 11 years
  Immunological assessments of peripheral blood mononuclear cells, serum and tissue biopsies (if any) will be reported using units appropriate to each particular assay. Results from immunohistochemical evaluations of tissue biopsies will be reported descriptively. Descriptive statistics will be used to summarize immunological findings. Any correlation with clinical response rate will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Butler, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada